CLINICAL TRIAL: NCT05595213
Title: Pilot Evaluation of Wrist Cooling Devices on the Severity of Hot Flashes for Women and Men Who Suffer From Moderate and or Severe Hot Flashes
Brief Title: Wrist Cooling for Hot Flashes Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-43277
Record Dates: First submitted 2022-10-21; First posted 2022-10-26 (Actual); Results first posted 2025-12-01 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Hot Flashes
Keywords: Breast cancer; Prostate cancer; Hormone deprivation therapy; Wrist cooling device
MeSH Terms: conditions — Hot Flashes; Breast Neoplasms; Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: In this study all participants will wear both the active wrist cooling device and the placebo device that look identical. However, the order that they wear the devices [which one they wear first or second] will be determined randomly.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Wrist Active Cooling and Placebo Device (Experimental): Each participant will be provided with two wrist devices [an active cooling device and a placebo device] that they will wear for 2 weeks each and during that time record the number of hot flashes in a study diary. The devices are worn like watches and that look identical. The order that they wear the devices will be randomly determined so some participants will wear the active cooling device first and then the placebo device and others will wear the placebo device first and then the active cooling device.
  Interventions: Device: Active cooling device with cooling plate; Device: Placebo device without cooling plate; Other: Hot Flash Diary

INTERVENTIONS:
Device: Active cooling device with cooling plate — This device is worn like a watch and pressing the button activates the cooling function to begin to cool the wrist skin temperature to 47 degrees. Pushing the device button again cools the skin to 60 degrees and a third time to 77degrees.
Device: Placebo device without cooling plate — This device is worn like a watch and pressing the button activates the cooling fan for 5 minutes.
Other: Hot Flash Diary — Participants will be instructed to document each hot flash experience daily and indicate if it was mild, moderate, or severe and whether they activated the wrist cooling device.

SUMMARY:
This pilot study aims to determine the impact of an experimental active cooling wrist device compared to a placebo device [the devices look identical] on symptom control of hot flashes in adult men and adult women experiencing hot flashes. The participants will record during the first two weeks of the study all of their hot flashes and severity of their hot flashes in a study diary. Each participant will wear each of the two devices [active cooling and placebo] during the trial but the order of which device they wear first will be determined by their random assignment into a group. The devices are identical in appearance and neither the participant nor the investigators w ill know which device the participants are wearing. Participants will wear the first assigned device for weeks 3 and 4. They will record in their diary the severity of their hot flashes while using the device. For weeks 5 and 6 they will use a second device and record in their diary the severity of their hot flashes with the use of the device.

The devices will be attached to the wrist like a watch. When activated, the experimental active cooling device will turn on a cooling fan with the cooling plate being active for up to 5 minutes. In contrast, the placebo device will only turn on a cooling fan for up to 5 minutes without the cooling plate being active.

ELIGIBILITY:
Inclusion Criteria:

1. Experiencing at least 2 hot flashes per day that are either moderate and/or severe in severity.

   1. Moderate: sensation of heat with sweating/dampness but able to continue activity with only brief fanning needed
   2. Severe: sensation of intense heat with sweating and causing disruption of current activity
2. English speaking

Exclusion Criteria:

1. Temperature sensitivity due to cooling associated with an autoimmune or vascular disorder, such as Raynaud's phenomena, peripheral arterial disease or any other reasons.
2. Any wrist skin sensitivity that is known to cause discomfort when any type of device such as a wristwatch is placed on the wrist.
3. Any lack of sensitivity to coolness on the wrists or hands
4. Any use of pharmaceuticals or devices to treat hot flashes.
5. Unable to understand and speak English

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2023-03-05 (Actual); Primary Completion 2025-01-02 (Actual); Study Completion 2025-01-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael F Holick, PhD MD, Principal Investigator — BU School of Medicine, Endocrinology
Locations (1):
- BU School of Medicine, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants recorded baseline frequency and severity for 2 weeks and then were randomly assigned the order of which of the two devices they would wear first [active cooling or placebo] which they did for 2 weeks. After 2 weeks of follow up they wore the other device for 2 weeks.
Groups:
- Used Active Cooling Device, Then Placebo Device: The active cooling wrist device was used for 2 weeks and after 2 weeks of follow-up the placebo device was used by each participant.
- Used Placebo Device, Then Active Cooling Device: The placebo device was used for 2 weeks and after 2 weeks of follow-up the active cooling device was used by each participant.
Period: Overall Study
Arm/Group | Used Active Cooling Device, Then Placebo Device | Used Placebo Device, Then Active Cooling Device
Started | 12 | 15
Completed | 12 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Wrist Active Cooling and Placebo Device: All participants wore both the active cooling and placebo devices for 2 weeks each. The order of which device was worn first was randomly determined.
Arm/Group | Wrist Active Cooling and Placebo Device
Number analyzed (Participants) | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.6 (15.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 12
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 27
Baseline number and severity of hot flashes [Number; unit: number of hot flashes]
  Mild | 785
  Moderate | 1317
  Severe | 1195

OUTCOME MEASURES:

1. Primary Outcome: Number and Severity of Hot Flashes
Description: Severity of hot flashes is defined as mild, moderate, and severe. The number of hot flashes by severity category are abstracted from the study 'hot flash diary'.
Time Frame: 6 weeks
Population: Each participant wore an active cooling wrist device and a placebo wrist device during the study so there are data on both for each of the 27 participants.
Measure: Number; unit: number of hot flashes
Groups:
- Active Cooling Device: This device is worn like a watch and pressing the button activates the cooling function to begin to cool the wrist skin temperature to 47 degrees. Pushing the device button again cools the skin to 60 degrees and a third time to 77degrees.
- Placebo Device: The placebo device device has the same porcelain plate that the cooling device has but it is not activated to cool when the device is turned on. This device is worn like a watch and pressing the button activates the fan for 5 minutes.
Arm/Group | Active Cooling Device | Placebo Device
Number analyzed (Participants) | 27 | 27
number of hot flashes
  Mild | 1148 | 692
  Moderate | 924 | 1213
  Severe | 633 | 1117

ADVERSE EVENTS:
Time Frame: 6 weeks
Groups:
- Active Cooling Device, Then Placebo Device: The active cooling wrist device was used for 2 weeks and after 2 weeks of follow-up the placebo device was used by each participant.
- Placebo Device, Then Active Cooling Device: The placebo device was used for 2 weeks and after 2 weeks of follow-up the active cooling device was used by each participant.
Arm/Group | Active Cooling Device, Then Placebo Device | Placebo Device, Then Active Cooling Device
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/27
Other Adverse Events (participants affected / at risk) | 0/27 | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-01-23): https://cdn.clinicaltrials.gov/large-docs/13/NCT05595213/Prot_SAP_000.pdf